CLINICAL TRIAL: NCT00345761
Title: Phase I/II Study of R340 (Capecitabine), L-OHP (Oxaliplatin) and R435 (Bevacizumab) in Advanced and/or Metastatic Colorectal Cancer
Brief Title: Clinical Study of Capecitabine, Oxaliplatin and Bevacizumab in Colorectal Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Chugai Pharmaceutical (Industry)
Collaborators: Yakult Honsha Co., LTD (Industry)
Responsible Party: Chugai Pharmaceutical CO.,LTD, Chugai Pharmaceutical CO.,LTD
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JO19380
Record Dates: First submitted 2006-06-27; First posted 2006-06-28 (Estimated); Last update posted 2010-08-16 (Estimated); Status verified 2010-08

CONDITIONS: Colorectal Cancer
Keywords: Advanced and/or metastatic colorectal cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Bevacizumab; Oxaliplatin; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Step 1 (Experimental)
  Interventions: Drug: Oxaliplatin; Drug: Capecitabine
- Step 2 (Experimental)
  Interventions: Drug: Bevacizumab; Drug: Oxaliplatin; Drug: Capecitabine
- Step 3 (Experimental)
  Interventions: Drug: Bevacizumab; Drug: Oxaliplatin; Drug: Capecitabine

INTERVENTIONS:
Drug: Bevacizumab — 7.5 mg/kg(i.v.) on Day 1 of 1 cycle(3 weeks)
  Arms: Step 2; Step 3
Drug: Oxaliplatin — 130 mg/m2(i.v.) on Day 1 of 1 cycle(3 weeks)
Drug: Capecitabine — 2000 mg/m2/day(p.o.) for 14 days in 1 cycle(3 weeks)

SUMMARY:
This study will evaluate the efficacy, safety and pharmacokinetics of capecitabine (2000 mg/m2/day by mouth [po], day 1 pm-day 15 am every 3 weeks [q3w]), oxaliplatin (130 mg/m2 intravenously [iv], day 1 q3w) and bevacizumab (7.5 mg/kg iv, day 1 q3w) in patients with advanced and/or metastatic colorectal cancer.

DETAILED DESCRIPTION:
This study will evaluate the efficacy, safety and pharmacokinetics of Capecitabine (2000 mg/m2/day po, day 1 pm-day 15 am q3w), Oxaliplatin (130 mg/m2 iv, day 1 q3w) and Bevacizumab (7.5 mg/kg iv, day 1 q3w) in patients with advanced and/or metastatic colorectal cancer.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients 20-74 years of age
* Histologically confirmed colorectal cancer
* Metastatic and/or locally advanced colorectal cancer not previously treated with chemotherapy for metastatic disease
* At least one measurable lesion according to RECIST

Exclusion Criteria:

* Evidence of clinically detectable ascites at study treatment start
* Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to study treatment start, or anticipation of the need for major surgical procedure during the course of the study; fine needle aspiration within 7 days prior to study treatment start.
* Evidence of bleeding diathesis or coagulopathy
* Serious, non-healing wound, ulcer, or bone fracture
* Chronic, daily aspirin (> 325 mg/day), anticoagulants, or other medications known to predispose to gastrointestinal ulceration

Ages: 20 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2006-02; Primary Completion 2008-10 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Response rate: Response Evaluation Criteria in Solid Tumors (RECIST) | event driven
Safety (Common Terminology Criteria for Adverse Events [CTCAE] version 3.0) | throughout study

SECONDARY OUTCOMES:
time to progression | event driven
overall survival | event driven
time to response | event driven
duration of response | event driven
concentrations of R340 and its metabolites | throughout study
concentrations of platinum | throughout study
concentrations of bevacizumab | throughout study
concentrations of vascular endothelial growth factor (VEGF) | throughout study
concentrations of anti-bevacizumab antibody | throughout study

CONTACTS AND LOCATIONS:
Overall Officials: Yuji Hayashi, Study Chair — Clinical Development Department 3, Group 6
Locations (4):
- Japan (4):
  - Hokkaido Region, Hokkaido, Hokkaido
  - Kanto Region, Kanto, Kanto
  - Kinki Region, Kinki, Kinki
  - Tokai Region, Tōkai, Tokai